CLINICAL TRIAL: NCT01586624
Title: A Cancer Research UK Phase I Dose Escalation Trial of Oral VEGFR and EGFR Inhibitor, Vandetanib in Combination With the Oral MEK Inhibitor, Selumetinib (VanSel-1) in Solid Tumours (Dose Escalation) and NSCLC (Expansion Cohort).
Brief Title: A Phase I Trial of Vandetanib (AZD6474) and Selumetinib (AZD6244) for Solid Tumours Including Non Small Cell Lung Cancer (VanSel-1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/11/001; 2011-000627-33 (EudraCT Number)
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Cancer; Non Small Cell Lung Cancer
Keywords: Phase I; Drug evaluation; Oncology; Vandetanib; Selumetinib; Dose escalation; Clinical trial; Vascular Endothelial Growth Factor (VEGFR) inhibitor; Epidermal Growth Factor Receptor (EGFR) inhibitor; Mitogen Activated Kinase (MEK) inhibitor; Non small cell lung cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Dose Escalation Phase Cohort 1 (Steady state dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) (Experimental): Dose escalation to determine recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Interventions: Drug: Vandetanib, Selumetinib
- Dose Escalation Phase Cohort 2 (Steady state dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) (Experimental): Dose escalation to determine recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Interventions: Drug: Vandetanib, Selumetinib
- Dose Escalation Phase Cohort 3 (Steady state dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) (Experimental): Dose escalation to determine recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Interventions: Drug: Vandetanib, Selumetinib
- Dose Escalation Phase Cohort 4 (Steady state dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) (Experimental): Dose escalation to determine recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Interventions: Drug: Vandetanib, Selumetinib
- Dose Escalation Phase Cohort 5a (Steady state dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) (Experimental): Dose escalation to determine recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Interventions: Drug: Vandetanib, Selumetinib
- Dose Escalation Phase Cohort 5b (Steady state dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) (Experimental): Dose escalation to determine recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Interventions: Drug: Vandetanib, Selumetinib
- Dose Escalation Phase Cohort 6 (Steady state dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib) (Experimental): Dose escalation to determine recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Interventions: Drug: Vandetanib, Selumetinib
- Expansion Phase (Steady state dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) (Experimental): Expansion cohort at the recommended phase 2 dose of vandetanib and selumetinib defined in the escalation phase.
  Interventions: Drug: Vandetanib, Selumetinib

INTERVENTIONS:
Drug: Vandetanib, Selumetinib — Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 25 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 25 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
  Arms: Dose Escalation Phase Cohort 1 (Steady state dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib)
Drug: Vandetanib, Selumetinib — Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
  Arms: Dose Escalation Phase Cohort 2 (Steady state dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib)
Drug: Vandetanib, Selumetinib — Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 75 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 75 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
  Arms: Dose Escalation Phase Cohort 3 (Steady state dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib)
Drug: Vandetanib, Selumetinib — Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 100 mg of selumetinib OD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 100 mg of selumetinib OD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
  Arms: Dose Escalation Phase Cohort 4 (Steady state dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib)
Drug: Vandetanib, Selumetinib — Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 125 mg of selumetinib OD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 125 mg of selumetinib OD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
  Arms: Dose Escalation Phase Cohort 5a (Steady state dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib)
Drug: Vandetanib, Selumetinib — Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 200 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
  Arms: Dose Escalation Phase Cohort 5b (Steady state dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)
Drug: Vandetanib, Selumetinib — Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 2) followed by vandetanib steady state dose of 300 mg OD (Days 3 to 14) followed by vandetanib steady state dose of 300 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 300 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
  Arms: Dose Escalation Phase Cohort 6 (Steady state dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib)
Drug: Vandetanib, Selumetinib — Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 200 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
  Arms: Expansion Phase (Steady state dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)

SUMMARY:
The purpose of this study is to determine whether using two drugs together called vandetanib and selumetinib is effective in the treatment of cancer. The first part of this study will include patients with any solid tumour and the second part of this study will include only patients with non small cell lung cancer. The four main aims of this clinical study are to find out:

* If the two drugs can be given safely to patients when given together.
* The maximum dose that can be given safely to patients.
* More about the potential side effects of the drugs and how they can be managed.
* What happens to vandetanib and selumetinib inside the body.

DETAILED DESCRIPTION:
The purpose of this Phase I study is to establish a safety and toxicity profile of combining two study drugs; vandetanib, a VEGFR (Vascular Endothelial Growth Factor Receptor) and EGFR (Epidermal Growth Factor Receptor) inhibitor, with selumetinib a MEK (Mitogen Activated Kinase) inhibitor.

This is the first time the drugs have been used together. These types of drugs have shown an effect in non small cell lung cancer (NSCLC).

The study is in two parts; the dose escalation phase and the expansion phase.

In the dose escalation phase, 42-50 patients will receive different doses of vandetanib and increasing doses of selumetinib to establish a safe dose to recommend for the next stage of the study. Patients with any solid tumour will be eligible.

In the expansion phase, up to 30 patients will receive the dose recommended in the previous phase. Only patients with NSCLC will be eligible for this part of the study.

The expansion phase will look at further evaluating the safety of the drug combination and the anti-tumour activity. Patients in this cohort will be requested to also consent to have additional imaging assessments and optional tumour biopsies.

Study treatment is administered orally; vandetanib tablets once daily and selumetinib capsules once daily (OD)/twice daily (BD). Cycle 1 is 42 days long. Subsequent cycles are 28 days in length. Patients will receive a total of 6 cycles of the combination treatment. If the patient has not progressed after six cycles, they may be treated for further cycles following approval from the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. (Dose escalation cohorts) Histologically or cytologically proven solid tumour for which no conventional therapy exists or is declined by the patient
2. (Expansion cohort only) Histologically or cytologically confirmed NSCLC patients only, for which no conventional therapy exists or is declined by the patient.

   * If only cytologically confirmed, baseline biopsy is mandatory for a patient to be eligible.
   * For NSCLC patients to be eligible for the expansion cohort they must have received:

     * One prior line of chemotherapy and/or
     * Previous platinum based chemotherapy and/or
     * At least one previous EGFR inhibitor
3. (Expansion cohort only) Measurable disease according to RECIST criteria Version 1.1 in final version of the protocol
4. Life expectancy of at least 12 weeks
5. World Health Organisation (WHO) performance status of 0-1
6. Baseline LVEF > 50%
7. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day -1) before the patient goes on study.

   Laboratory Test Value required

   Haemoglobin (Hb) ≥ 9.0 g/dL

   Absolute neutrophil count ≥ 1.5 x 10^9/L

   Platelet count ≥ 100 x 10^9 /L

   Normal serum calcium (adjusted)* 2.15-2.55 mmol/L

   Normal serum magnesium* 0.60-1.0 mmol/L

   Normal serum potassium >4.0 mmol/L

   Either: Serum bilirubin ≥1.5 x upper limit of normal (ULN) This does not apply to patients with Gilbert's disease.

   Alanine amino-transferase (ALT) or aspartate amino-transferase (AST) and alkaline phosphatase (ALP) ≤ 2.5 x ULN unless raised due to liver metastases in which case up to 5 x ULN is permissible

   Either: Calculated creatinine clearance (using the Wright or C&G formula) > 50 mL/min

   Or: Isotope clearance measurement** ≥ 50 mL/min (uncorrected)

   INR or aPTT < 1.5 x ULN

   *or normal range according to the local laboratory

   ** Isotope clearance result to be used to confirm eligibility if calculated C&G/Wright method results in GFR of = 50 mL/min.

   *** Therapeutic INR values (2.0-3.0) are acceptable to confirm eligibility for patients who are taking concomitant warfarin.
8. 18 years or over
9. Ability to swallow and retain oral medications.
10. Written (signed and dated) informed consent and be capable of co-operating with treatment, and follow-up

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous 4 weeks (6 weeks for investigational medicinal products) before treatment.
2. Patients who have been withdrawn from treatment with agents that target EGFR because of unacceptable toxicity (prior treatment with these agents is allowed) and those patients who have had EGFR dose reductions by 50% or more.
3. Expansion cohort only: Prior treatment with any agent that targets MEK or VEGFR
4. Any prior exposure to RAS or RAF inhibitors
5. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 2 toxicities, which in the opinion of the Investigator and the Centre for Drug Development (CDD) should not exclude the patient.
6. Symptomatic brain metastases (patients must be stable for >3 months post RT treatment) or spinal cord compression.
7. Patients with interstitial lung disease.
8. Pregnant or lactating women are excluded. Female patients with the ability to become pregnant who have a negative serum or urine pregnancy test before enrollment and agree to use two of the following three highly effective forms of combined contraception (oral, injected or implanted hormonal contraception and condom, have a intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.
9. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (e.g. condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
10. Major surgery from which the patient has not yet recovered.
11. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
12. Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
13. Cardiac conditions as follows:

    * Clinically significant cardiovascular event within 3 months prior to entry to include:

      * Myocardial infarction
      * Angina requiring use of nitrates more than once weekly
      * Superior vena cava syndrome
      * Class II/III/IV cardiac disease (New York Heart Association [NYHA])
      * Presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
    * History of arrhythmia which is symptomatic or requires treatment (CTCAE V4.02), symptomatic or uncontrolled atrial fibrillation despite treatment or asymptomatic sustained ventricular tachycardia. Patients with atrial fibrillation controlled by medication are permitted.
    * Uncontrolled hypertension (BP > 160/100 despite optimal therapy)
    * Prior or current cardiomyopathy
    * Atrial fibrillation with heart rate > 100 bpm
    * QTcB > or equal to 450 msec on screening ECG (Note: If a patient has a QTcB interval > or equal to 450 msec on screening ECG, the screen ECG may be repeated twice [at least 24 hours apart]. The average QTcB from the three screening ECGs must be < 450 msec in order for the subject to be eligible for the study.)
    * History of congenital long QT syndrome
    * History of Torsade de Pointes (or any concurrent medication with a known risk of inducing Torsades de Pointes.)
14. Concomitant medications that are potent inducers of CYP3A4 function i.e. rifampicin, rifabutin, phenytoin, carbamazepine, Phenobarbital and St John"s Wort.
15. Any other condition which in the Investigator"s opinion would not make the patient a good candidate for the clinical trial (e.g. evidence of severe or uncontrolled systemic disease or concurrent condition or that may affect ability to absorb oral agents).
16. Current malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for five years or more and are deemed at negligible risk for recurrence, are eligible for the trial.
17. If a participant plans to participate in another interventional clinical study, whilst taking part in this Phase I study. Participation in an observational study would be acceptable.
18. Ophthalmological conditions as follows:

    1. Current or past history of retinal pigment epithelial detachment (RPED)/central serous retinopathy (CSR) or retinal vein occlusion.
    2. Intraocular pressure (IOP) > 21 mmHg or uncontrolled glaucoma (irrespective of IOP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Talbot, Prof, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (4):
- United Kingdom (4):
  - Churchill Hospital, Headington, Oxford
  - Addenbrooke's Hospital, Cambridge
  - The Christie Hospital, Manchester
  - Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Simple summary of trial results on Cancer Research UK Trial Database — https://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-of-vandetanib-and-selumetinib-for-solid-tumours-including-nsclc-vansel-1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial participants were enrolled at three trial sites between 10 January 2012 and 19 September 2017.
Groups:
- Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 25 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 25 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 75 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 75 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 100 mg of selumetinib OD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 100 mg of selumetinib OD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 125 mg of selumetinib OD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 125 mg of selumetinib OD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 200 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 2) followed by vandetanib steady state dose of 300 mg OD (Days 3 to 14) followed by vandetanib steady state dose of 300 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 300 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib): Expansion cohort at the recommended phase 2 dose of vandetanib and selumetinib defined in the escalation phase.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 200 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
Period: Overall Study
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)
Started | 6 | 6 | 6 | 7 | 9 | 8 | 8 | 11
Completed | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Not Completed | 4 | 4 | 5 | 7 | 8 | 8 | 8 | 10
Not completed — Adverse Event | 3 | 0 | 2 | 1 | 3 | 3 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Evidence of disease progression | 1 | 3 | 2 | 5 | 3 | 5 | 4 | 6
Not completed — Screen failure (no treatment received) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib ): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib ): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 75 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 75 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 2) followed by vandetanib steady state dose of 300 mg OD (Days 3 to 14) followed by vandetanib steady state dose of 300 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 300 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib): Expansion cohort at the recommended phase 2 dose of vandetanib and selumetinib defined in the escalation phase.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 200 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 200 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib ) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib ) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib) | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 9 | 8 | 8 | 11 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 3 | 5 | 3 | 3 | 4 | 6 | 29
  >=65 years | 6 | 1 | 3 | 2 | 6 | 5 | 4 | 5 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 4 | 2 | 6 | 4 | 6 | 31
  Male | 3 | 4 | 2 | 3 | 7 | 2 | 4 | 5 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 7 | 9 | 8 | 8 | 11 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events, Non-serious Adverse Events and Treatment Emergent Adverse Events.
Description: Number of serious adverse events, non-serious adverse events and treatment emergent adverse events.
Time Frame: Safety data was collected from the date of written informed consent and continued until 28 days after the final administration of vandetanib and selumetinib, an average (mean) of 164 days (approximately 5.4 months).
Population: All patients who met the eligibility criteria and received at least one dose of the combination treatment (vandetanib and selumetinib) were evaluable for safety assessment (N=57).
Measure: Number; unit: Adverse events
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib) | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 8 | 7 | 6 | 11
Adverse events
  Total SAEs | 10 | 11 | 13 | 5 | 28 | 10 | 14 | 14
  Total NSAEs | 99 | 90 | 70 | 94 | 161 | 98 | 114 | 130
  Total treatment emergent AEs | 107 | 99 | 79 | 93 | 165 | 102 | 126 | 135

2. Primary Outcome: Number of Dose Limiting Toxicities (DLTs) Within Each Cohort.
Description: Number of DLTs within each cohort.
Time Frame: DLTs occurring in the first Cycle (up to Day 42).
Population: as for outcome 1
Measure: Number; unit: DLTs
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib) | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 8 | 7 | 6 | 11
DLTs | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 2

3. Secondary Outcome: Dose Escalation Cohorts Only: PK Parameter Maximum Observed Plasma Concentration of Vandetanib.
Description: Maximum observed plasma concentration of vandetanib post treatment with vandetanib alone and following the combination of vandetanib and selumetinib.
Time Frame: 0 hours (pre dose) and at 0.5, 2, 4, 6 and 24 hours post dose on Day 4. 0 hours (pre dose) and at 0.5, 2, 4, 6, 10 and 24 hours post dose on Days 15 and 29.
Population: All patients in the dose escalation cohorts (Cohorts 1 to 6) who received at least one dose of IMP (N=47 with available PK data).
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 8 | 8 | 6
ng/mL
  Day 4 | 585 [428 to 947] | 561 [223 to 1500] | 582 [422 to 890] | 790 [337 to 1210] | 484.5 [379 to 733] | 702.5 [382 to 910] | 702 [526 to 1390]
  Day 15 | 503.5 [319 to 765] | 436 [206 to 703] | 414.5 [367 to 605] | 476 [301 to 796] | 401.5 [273 to 592] | 701 [446 to 1260] | 906 [713 to 1380]
  Day 29 | 556 [384 to 690] | 399 [284 to 605] | 538 [288 to 704] | 503 [306 to 695] | 335.5 [183 to 346] | 988 [522 to 1240] | 902 [481 to 1160]

4. Secondary Outcome: Dose Escalation Cohorts Only: PK Parameter Maximum Observed Plasma Concentration of Selumetinib.
Description: Maximum observed plasma concentration of selumetinib post treatment with the combination of vandetanib and selumetinib.
Time Frame: 0 hours (pre dose) and at 0.5, 2, 4, 6, 10 and 24 hours post dose on Days 15 and 29.
Population: as for outcome 3
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 8 | 8 | 6
ng/mL
  Day 15 | 324.5 [134 to 698] | 605 [415 to 828] | 1280 [529 to 1870] | 1890 [320 to 3060] | 2005 [853 to 2810] | 501 [326 to 782] | 814 [489 to 981]
  Day 29 | 430 [193 to 852] | 569 [363 to 1030] | 1220 [553 to 1920] | 1740 [1370 to 2550] | 1440 [1430 to 2190] | 587 [564 to 1200] | 593 [262 to 1100]

5. Secondary Outcome: Dose Escalation Cohorts Only: PK Parameter Area Under the Plasma Concentration Time Curve (0-24 Hours) of Vandetanib.
Description: Area under the plasma concentration time curve (0-24 hours) of vandetanib post treatment with vandetanib alone and following the combination of vandetanib and selumetinib.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 8 | 8 | 6
h*ng/mL
  Day 4 | 12032 [9115 to 19402] | 11629.5 [4861 to 30192] | 11189 [8989 to 17979] | 16603 [7448 to 21877] | 10286.5 [8056 to 14169] | 14395 [8082 to 20965] | 14830.5 [11310 to 26269]
  Day 15 | 9253.5 [6583 to 15931] | 8822.5 [4659 to 15225] | 7958.5 [7047 to 13606] | 9946 [6142 to 17340] | 8814.5 [6045 to 13325] | 15442 [8212 to 27375] | 18864 [14032 to 29896]
  Day 29 | 12555 [8673 to 15077] | 8355 [5977 to 13598] | 11246 [6434 to 15271] | 10058 [6871 to 15763] | 7261.5 [3801 to 7482] | 18573 [11362 to 25692] | 15923 [9987 to 24112]

6. Secondary Outcome: Dose Escalation Cohorts Only: PK Parameter Area Under the Plasma Concentration Time Curve (0-12 Hours) of Selumetinib.
Description: Area under the plasma concentration time curve (0-12 hours) of selumetinib post treatment with the combination of vandetanib and selumetinib. This was extrapolated from the sampling data up to 10 hours to allow comparison with literature data.
Time Frame: 0 hours (pre dose) and at 0.5, 2, 4, 6 and 10 hours post dose on Days 15 and 29.
Population: as for outcome 3
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 8 | 8 | 6
h*ng/mL
  Day 15 | 1251.5 [639 to 2361] | 2050 [1542 to 3607] | 4072.5 [2111 to 5615] | 6138 [2045 to 10777] | 6921 [4600 to 9329] | 1698 [1391 to 3028] | 2770 [2015 to 3550]
  Day 29 | 1913 [1400 to 2122] | 2550 [1386 to 4494] | 4762 [2685 to 9798] | 6998 [4165 to 11326] | 6429 [6306 to 7768] | 3049 [2843 to 3753] | 2477 [1094 to 3277]

7. Secondary Outcome: Dose Escalation Cohorts Only: PK Parameter Area Under the Plasma Concentration Time Curve (0-12 Hours) of N-desmethyl Metabolite of Selumetinib.
Description: Area under the plasma concentration time curve (0-12 hours) of N-desmethyl metabolite of selumetinib following the combination of vandetanib and selumetinib. This was extrapolated from the sampling data up to 10 hours to allow comparison with literature data.
Time Frame: 0 hours (pre dose) and at 0.5, 2, 4, 6 and 10 hours post dose on Days 15 and 29.
Population: as for outcome 3
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 (Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 8 | 8 | 6
h*ng/mL
  Day 15 | 78.5 [44 to 149] | 141 [127 to 332] | 255 [88 to 407] | 349 [145 to 925] | 493 [328 to 686] | 182 [95 to 338] | 236 [144 to 340]
  Day 29 | 89 [59 to 251] | 163 [126 to 288] | 230 [125 to 535] | 390 [189 to 758] | 377 [348 to 383] | 293 [173 to 475] | 205 [83 to 256]

8. Secondary Outcome: Expansion Cohort Only: Progression Free Survival (PFS) of Patients With NSCLC After Treatment With the Combination of Vandetanib and Selumetinib.
Description: PFS by Response Evaluation Criteria in Solid Tumours Criteria (RECIST v1.0). Per RECIST for target lesions and assessed by computerised tomography (CT), progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum while on trial, or the appearance of one or more new lesions.
Time Frame: 10 and 18 weeks from date of first dose of vandetanib.
Population: All patients in the expansion cohort receiving at least one cycle* of the vandetanib and selumetinib combination with a baseline assessment of disease (N=9).
  *To be evaluable for response, a patient must have received a minimum of 21 of the 28 daily doses of the combination treatment in Cycle 1.
Measure: Number; unit: participants
Arm/Group | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 9
participants
  Progression free at 10 weeks | 3
  Progression free at 18 weeks | 2

9. Secondary Outcome: Expansion Cohort Only: One Year Survival of Patients With NSCLC After Treatment With the Combination of Vandetanib and Selumetinib.
Description: Number of patients alive at one year.
Time Frame: 1 year from date of first dose of vandetanib.
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 9
participants | 2

10. Secondary Outcome: Expansion Cohort Only: Tumour Metabolism in Patients With NSCLC Using Positron Emission Tomography Response Criteria in Solid Tumours (PERCIST) Criteria.
Description: Tumour metabolism using 18F-fluorodeoxyglucose positron emission tomography ([18F]FDG-PET) computerised tomography (CT) imaging pre and post treatment with vandetanib alone and following the combination of vandetanib and selumetinib. These were assessed and reported according to PERCIST criteria.
Time Frame: Baseline, Day 12, Day 42.
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)
Number analyzed (Participants) | 9
participants
  Day 12 Complete Metabolic Response | 0
  Day 12 Partial Metabolic Response | 0
  Day 12 Stable Metabolic Disease | 8
  Day 12 Progressive Metabolic Disease | 1
  Day 42 Complete Metabolic Response | 0
  Day 42 Partial Metabolic Response | 2
  Day 42 Stable Metabolic Disease | 3
  Day 42 Progressive Metabolic Disease | 2
  Day 42 Not assessed | 2

ADVERSE EVENTS:
Time Frame: Safety data was collected from the date of written informed consent and continued until 28 days after the final administration of vandetanib and selumetinib, an average (mean) of 164 days (approximately 5.4 months). Overall Mortality was collected during the Safety data assessment period for the dose Escalation Cohorts and up to one year after Cycle 1 Day 1 for the Expansion Cohort.
Description: Per protocol, where deaths due to disease progression were reported as AEs, these weren't considered to be SAEs unless related to the IMP. These events were coded by the Sponsor as "Death NOS" in the clinical database but have been entered as disease progression at the request of ClinicalTrials.gov. For patients recruited to the expansion cohort, deaths due to disease progression in the survival follow-up period were not reported as AEs but have been included in the All-cause mortality numbers.
Groups:
- Dose Escalation Phase Cohort 2 ( Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib): Dose escalation to determine the recommended dose and schedule for Phase 2 evaluation of vandetanib and selumetinib.
  Cycle 1: Vandetanib higher (lead in) dose of 300 mg OD (Days 1 to 4) followed by vandetanib steady state dose of 100 mg OD (Days 5 to 14) followed by vandetanib steady state dose of 100 mg OD + 50 mg of selumetinib BD (28 days). Cycle 1 is 42 days long.
  Cycle 2 onwards: Vandetanib steady state dose of 100 mg OD + 50 mg of selumetinib BD (28 days). From Cycle 2, cycles are 28 days long.
  Patients will be allowed to receive 6 cycles. If the patient is still benefiting clinically with no unacceptable toxicity, then the Investigator can ask the Sponsor for continuation of treatment.
Arm/Group | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) | Dose Escalation Phase Cohort 2 ( Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib) | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/6 | 2/6 | 0/7 | 1/8 | 0/7 | 1/6 | 7/11
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/6 | 6/6 | 2/7 | 7/8 | 5/7 | 6/6 | 8/11
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 7/7 | 8/8 | 7/7 | 6/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) (N=6) | Dose Escalation Phase Cohort 2 ( Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) (N=6) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) (N=6) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) (N=7) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) (N=8) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) (N=7) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib) (N=6) | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) (N=11)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 1 (1)
Retinal detachment (Eye disorders) | 0 | 0 | 2 (2) | 0 | 3 (4) | 1 (1) | 3 (3) | 1 (1)
Retinal vascular disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Retinopathy (Eye disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 1 (3) | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 | 2 (8) | 0 | 1 (2) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 1 (4) | 0 | 0 | 1 (1)
Disease Progression (General disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Lung infection (Infections and infestations) | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Stroke (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2)
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 3 (3) | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 3 (3)
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase Cohort 1 (Steady State Dose of 100 mg OD Vandetanib + 25 mg BD Selumetinib) (N=6) | Dose Escalation Phase Cohort 2 ( Steady State Dose of 100 mg OD Vandetanib + 50 mg BD Selumetinib) (N=6) | Dose Escalation Phase Cohort 3 (Steady State Dose of 100 mg OD Vandetanib + 75 mg BD Selumetinib) (N=6) | Dose Escalation Phase Cohort 4 (Steady State Dose of 100 mg OD Vandetanib + 100 mg OD Selumetinib) (N=7) | Dose Escalation Phase Cohort 5a (Steady State Dose of 100 mg OD Vandetanib + 125 mg OD Selumetinib) (N=8) | Dose Escalation Phase Cohort 5b (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) (N=7) | Dose Escalation Phase Cohort 6 (Steady State Dose of 300 mg OD Vandetanib + 50 mg BD Selumetinib) (N=6) | Expansion Phase (Steady State Dose of 200 mg OD Vandetanib + 50 mg BD Selumetinib) (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 0
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1 (1) | 0 | 1 (2) | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 | 0 | 2 (2) | 0 | 0 | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Blurred vision (Eye disorders) | 2 (2) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 | 0 | 0 | 2 (2) | 0 | 1 (1) | 0 | 1 (1)
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Flashing lights (Eye disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 | 0 | 1 (3) | 3 (6) | 3 (3) | 2 (2) | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (3) | 1 (1) | 2 (3) | 2 (3) | 2 (2) | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (7) | 5 (12) | 5 (6) | 4 (6) | 5 (17) | 7 (17) | 5 (14) | 8 (16)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 1 (3) | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 1 (3) | 0 | 0 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 | 1 (1) | 2 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (6) | 3 (5) | 5 (9) | 4 (8) | 4 (8) | 3 (6) | 4 (8)
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2)
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 (2) | 0 | 0 | 1 (1) | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (4) | 3 (4) | 5 (10) | 1 (4) | 4 (10) | 2 (4) | 2 (4)
Chills (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) — Death due to disease progression (not considered related to IMP). Per protocol, cases of death due to disease progression were not considered to be SAEs, unless considered related to the IMP.
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Fatigue (General disorders) | 3 (4) | 5 (5) | 5 (7) | 3 (4) | 3 (3) | 2 (2) | 2 (2) | 6 (10)
Fever (General disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1) | 0
Flu like symptoms (General disorders) | 1 (2) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 0 | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 0 | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Infections and infestations - Other, specify (Infections and infestations) | 3 (3) | 0 | 2 (3) | 1 (1) | 3 (4) | 1 (2) | 0 | 2 (4)
Lung infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 1 (2) | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2)
Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Paronychia (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2)
Skin infection (Infections and infestations) | 0 | 1 (1) | 1 (1) | 2 (3) | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (3) | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 | 2 (2) | 0 | 2 (2) | 2 (2) | 4 (5) | 2 (2)
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (2)
Cardiac troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Cholesterol high (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
CPK increased (Investigations) | 0 | 1 (1) | 2 (2) | 0 | 2 (3) | 0 | 3 (7) | 4 (6)
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 2 (2)
Ejection fraction decreased (Investigations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2) | 0 | 0 | 0 | 3 (3) | 2 (2) | 4 (7) | 0
Investigations - Other, specify (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (6) | 0
Weight loss (Investigations) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 | 3 (6) | 0 | 1 (1) | 1 (1) | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 1 (1) | 0 | 2 (6) | 1 (1) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 (2) | 1 (1) | 0 | 4 (7) | 1 (1) | 0 | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 | 0 | 2 (5) | 2 (2) | 0 | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 1 (2) | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 1 (3) | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 (2) | 0 | 1 (1) | 1 (3) | 0 | 1 (1) | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 (1) | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 2 (2) | 1 (1) | 0 | 1 (2) | 0 | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (2) | 0
Presyncope (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 | 0 | 3 (4) | 0 | 0 | 0
Libido increased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 | 2 (2) | 0 | 2 (2) | 2 (2) | 1 (1) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 2 (2) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1) | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 0 | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 (2) | 1 (1) | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 2 (2) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 | 3 (4) | 0 | 0 | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 1 (2) | 0 | 0 | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 | 1 (1) | 1 (1) | 3 (5) | 2 (3) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (7) | 3 (3) | 2 (4) | 4 (4) | 5 (7) | 3 (4) | 0 | 7 (8)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 3 (4) | 3 (4) | 5 (5)
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
61 patients were enrolled. 3 withdrew before having vandetanib (Van) or selumetinib (Sel). 1 patient in Cohort 5b received Van but withdrew before having Sel and was excluded from the safety analysis. The remaining 57 patients had at least 1 dose of the combination and were included in the safety analysis population (46 in dose escalation, 11 in expansion). PFS was planned to be assessed at 12 weeks but was instead assessed at 10 and 18 weeks as disease assessments were performed every 2 cycles

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT01586624/Prot_000.pdf